CLINICAL TRIAL: NCT02957201
Title: The Effect on Endothelial Progenitor Cells (EPCs) by Successful Cardiac Occlusion Device Implantation
Brief Title: The Effect on EPCs by Successful Cardiac Occlusion Device Implantation
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 997
Record Dates: First submitted 2016-10-20; First posted 2016-11-07 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2016-11

CONDITIONS: Foramen Ovale, Patent; Heart Septal Defects, Atrial; Atrial Septal Defect
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood samples (Other): Blood samples taken at baseline, day 1-2, day 3-4 and day 7-8 for Endothelial Progenitor Analysis with flow cytometer
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples at baseline and 3 timepoints for EPC analysis

SUMMARY:
All patients awaiting to have either a left atrial appendage closure (LAA) or patent foramen ovale (PFO) or Atrial Septal Defect (ASD) closure device as part of standard care will be identified and reviewed in cardiology clinics. These patients will be placed on waiting list to undergo the procedure. Patient-participants will be consented on the date of admission for device closure implantation.

The study will recruit 20 patients divided into; 10 patients undergoing PFO/ASD closure and 10 patients undergoing LAA closure. EPC will be measured on the day of the device implantation, day 0 and prior to discharge on day 1.

Patient participants are admitted overnight after the device closure implantation. Then on subsequent out patient cardiology research clinic follow appointments on days (3-4) and (7-8).

DETAILED DESCRIPTION:
The objective of this study is to assess the effect, if any, on EPC count and cardiac device implantation.

All patients awaiting LAA or PFO/ASD occlusion will firstly be reviewed in a cardiology clinic and assessed. Suitable patients will then be placed on a waiting list for occlusion device implantation and therefore identified as potential participants in the study. Patient-participants will be informed of the trial and given a chance to participate, this may be by face to face and or via invitation letter. All patient-participants will be given a copy of the patient information sheet.

Formal consent to participate in the trial will occur on the morning of the procedure. This will avoid repeated visits by patients that may have to travel some considerable distance.

The study will recruit 20 patients divided into; 10 patients undergoing PFO/ASD occlusion and 10 patients undergoing LAA occlusion. EPC will be measured on the day of the device implantation, day 0 and prior to discharge on day 1, then on subsequent follow up appointments on days (3-4) and (7-8). Blood samples of 3-5ml will be taken to allow flow cytometric analysis for EPCs.

Standard follow up for participants may include transesophageal echocardiography (TOE) at 3 months after implantation. This will give a direct assessment of device related thrombus. Currently TOE is not standard of care in PFO follow up. If a TOE result is available for either group the investigators will use the results in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over and suitable for cardiac device closure

Exclusion Criteria:

* Patients unable to give informed consent or attend follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Number of EPC cells per microliter of blood following cardiac closure device implantation | day 8
  Number of EPC cells per microliter of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Butler Robert, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No